CLINICAL TRIAL: NCT04156815
Title: Treatment of Acne Vulgaris Using 1,565 nm Non-ablative Fractional Laser in Combination With Isotretinoin and Pricking Blood Therapy
Brief Title: Treatment of Acne Vulgaris Using NAFL in Combination With Isotretinoin and Pricking Blood Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: xjpfW
Record Dates: First submitted 2019-10-09; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Acne scars; 1,565 nm non-ablative fractional laser; Isotretinoin; pricking blood therapy
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1,565nm NAFL only group (Active Comparator): Patients were first treated by the 1,565nm M22-ResurFx NAFL on inflammatory papules and boxcar atrophic scars using round or rectangle light spots with similar sizes of individual lesional papules or scars. The energy fluence was 60 mJ and spot density was 150 spots/cm2. A whole face pass treatment was followed using hexagon or rectangle light spots with fluences of 40-45 mJ, density of 200 spots/cm2 and no overlap on light spots. The end points of the treatment were appearance of localized erythema, edema and bruise on treated areas. A facial sheet mask (skin repair dressing, Panion & BF Biotech Inc, Zhuhai, China) was used to clean the face after laser treatment, and the face was cooled by air cooler for 10 minutes. The patients received three treatment sessions with a 6-week interval between each session.
  Interventions: Radiation: 1,565nm NAFL
- Oral isotretinoin only group (Active Comparator): Subjects received oral isotretinoin (Xingyi Yan'an Pharmaceutical, Shanghai, China) (1mg/kg/d for the first 2-4 weeks and 0.5mg/kg/d for the next 12-14 weeks) for a total of 16 weeks. Serum triglycerides, cholesterol and levels of liver enzymes were monitored every month during oral isotretinoin medication.
  Interventions: Drug: Oral isotretinoin
- Double therapy group (Active Comparator): The patients first received 2-4 weeks of oral isotretinoin medication (1mg/kg/d), followed by 1565nm M22-ResurFx NAFL treatment. Subjects were then given isotretinoin with a dosage of 0.5 mg/kg/d for the next 12-14 weeks. Laser treatment parameters and procedures were as same as in the group one above.
  Interventions: Radiation: 1,565nm NAFL; Drug: Oral isotretinoin
- Triple therapy group (Experimental): The patients received the same treatments as the subjects in group (3) with additional PBT. At the end point of each session of laser treatment, an acupuncture practitioner performed a PBT in the areas within 1.5 cm radius of the five facial acupoints (Yintang, Zhukong, Sun, Yingxiang, Cuanzhu) (Figure 1). These areas usually appeared intensive erythema. A facial sheet mask was used to clean the face after PBT, and the face was cooled by air cooler for 10 minutes.
  Interventions: Radiation: 1,565nm NAFL; Drug: Oral isotretinoin; Other: Pricking blood therapy

INTERVENTIONS:
Radiation: 1,565nm NAFL — 1,565nm M22-ResurFx NAFL can deliver additional benefits to existing acne scar and skin texture. Patients were first treated by the 1,565nm M22-ResurFx NAFL on inflammatory papules and boxcar atrophic scars using round or rectangle light spots with similar sizes of individual lesional papules or scars. The energy fluence was 60 mJ and spot density was 150 spots/cm2. A whole face pass treatment was followed using hexagon or rectangle light spots with fluences of 40-45 mJ, density of 200 spots/cm2 and no overlap on light spots. The end points of the treatment were appearance of localized erythema, edema and bruise on treated areas.
  Arms: 1,565nm NAFL only group; Double therapy group; Triple therapy group
Drug: Oral isotretinoin — Oral isotretinoin has remained the most effective medication for moderate-to-severe AV.Subjects received oral isotretinoin (Xingyi Yan'an Pharmaceutical, Shanghai, China) (1mg/kg/d for the first 2-4 weeks and 0.5mg/kg/d for the next 12-14 weeks) for a total of 16 weeks. Serum triglycerides, cholesterol and levels of liver enzymes were monitored every month during oral isotretinoin medication.
  Arms: Double therapy group; Oral isotretinoin only group; Triple therapy group
Other: Pricking blood therapy — Pricking blood therapy (PBT) is a modified acupuncture strategy that is adapted to treat inflammatory related diseases. It has been shown to be effective in treatment of many chronic and acute inflammatory conditions including vasomotor rhinitis, acute herpes zoster and acute gouty arthritis,suggesting a potential efficacy for AV as well. At the end point of each session of laser treatment, an acupuncture practitioner performed a PBT in the areas within 1.5 cm radius of the five facial acupoints (Yintang, Zhukong, Sun, Yingxiang, Cuanzhu) (Figure 1). These areas usually appeared intensive erythema. A facial sheet mask was used to clean the face after PBT, and the face was cooled by air cooler for 10 minutes.
  Arms: Triple therapy group

SUMMARY:
BACKGROUND Isotretinoin remains one of the first line medications for moderate-to-severe acne vulgaris (AV) but its side effect is a major concern for Asian patients.

OBJECTIVE Investigators aimed to evaluate the efficacy and safety of the 1,565 nm non-ablative fractional laser (NAFL) in combination with isotretinoin and pricking blood therapy (PBT) for treatment of AV.

METHODS A retrospective analysis of 60 patients with moderate-to-severe AV was performed. Four groups (n=15) were evaluated: 1,565nm NAFL alone, oral isotretinoin alone, double therapy (NAFL + isotretinoin) and triple therapy (NAFL + isotretinoin + PBT).

DETAILED DESCRIPTION:
BACKGROUND Isotretinoin remains one of the first line medications for moderate-to-severe acne vulgaris (AV) but its side effect is a major concern for Asian patients.

OBJECTIVE Investigators aimed to evaluate the efficacy and safety of the 1,565 nm non-ablative fractional laser (NAFL) in combination with isotretinoin and pricking blood therapy (PBT) for treatment of AV.

METHODS A retrospective analysis of 60 patients with moderate-to-severe AV was performed. Four groups (n=15) were evaluated: 1,565nm NAFL alone, oral isotretinoin alone, double therapy (1,565 nm non-ablative fractional laser + isotretinoin) and triple therapy (1,565 nm non-ablative fractional laser+ isotretinoin + PBT).

ELIGIBILITY:
Inclusion Criteria:

* Patients ranged in age from twenty to forty years old
* Clinically diagnosed as a facial acne patient
* The patients meet the needs of the research program of this topic

Exclusion Criteria:

* pregnancy
* liver or kidney functional abnormality
* skin ulceration with active bacteria
* fungal or viral infection or skin cancer
* coagulation disorders
* patients on drugs of agents
* systemic diseases such as cardiovascular disease
* epilepsy
* diabetes
* immunodeficiency disease
* active psoriasis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Visia CR imaging system | change from week0 to week24
  With fast capture times and lighting modes designed to enhance the visualization
Antera3D® system | change from week0 to week24
  The indexes of facial skin texture and other datas were quantitatively measured by the Antera3D® system before and after treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No